CLINICAL TRIAL: NCT00878085
Title: fMRI and Robot-Assisted Practice of Activities of Daily Living
Brief Title: Functional Magnetic Resonance Imaging (fMRI) and Robot-Assisted Practice of Activities of Daily Living
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Marquette University (Other)
Responsible Party: Principal Investigator, Michelle J. Johnson, Adjunct Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR; NIH 1K25NS058577 - 01A1
Record Dates: First submitted 2009-03-23; First posted 2009-04-08 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Hemiparesis; Ischemic Stroke; Chronic
Keywords: Robot Therapy; Upper Limb; Stroke; Rehabilitation; fMRI; DTI
MeSH Terms: conditions — Paresis; Ischemic Stroke; Bronchiolitis Obliterans Syndrome; Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Robot Therapy with activities of daily living (ADLs)
  Interventions: Device: Robot Therapy Device
- 2 (Active Comparator): Standard Occupational Therapy
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Device: Robot Therapy Device — 3x a week for 4 weeks
  Arms: 1
Behavioral: Occupational Therapy — 3x a week for 4 weeks
  Arms: 2

SUMMARY:
The investigators will study motor recovery after robot-assisted therapy after stroke. A small clinical trial will be conducted to quantify the central nervous system changes associated with robotic or standard training, and identify trends across high and low responders in terms of patterns of change in cortical activity and type of white matter connectivity.The investigators hypothesize that robot training will lead to larger improvements as compared to standard occupational therapy. The investigators hypothesize that high responders to the robot training will have reduced compensatory activation in the bilateral area and will connectivity in the motor tracts.

DETAILED DESCRIPTION:
Robot-assisted therapy is on the cutting edge of stroke rehabilitation and is a therapy method that promises to improve the lives of persons with disabilities due to stroke. Preliminary studies using these tools provide mixed evidence for their effectiveness and reveal limitations. For example, inconsistent carryover of motor gains to real life activities of daily living (ADLs) is seen. Therefore, it is still not clear what treatment strategies maximize functional outcomes on ADLs. There is a need to study the stroke recovery process and to understand how to optimize robot-assisted therapies in order to enhance patient rehabilitation and improve functional outcomes. Imaging techniques such as functional Magnetic Resonance Imaging (fMRI) and Diffusion Tensor Imaging (DTI) can assist us in understanding the stroke recovery process, in determining who may benefit from robot-assisted training, and in defining how training induced functional cortical changes occur after robot training. We propose to conduct an interventional study plus control to assess the effectiveness of four weeks of robot-assisted practice of tasks with skilled functional tasks that involve reaching and grasping activities similar to real activities. We will examine the process of recovery for low-to-moderate functioning stroke survivors with chronic disability. We will assess the ability of active-assisted reaching and grasping training to effect immediate gains and long-term functional improvements. Further, using fMRI and DTI, we plan to associate changes seen in motor impairment levels and functional task performance levels with white matter injuries and connectivity and changes in oxygen utilization in the motor cortex as well as other areas of the brain. Our short-term aims are to, i) assess short-term functional gains after practice of skilled reaching and grasping tasks; ii) assess maintenance of these improvements; iii) quantify the neuronal changes associated with short-term gains, and iv) identify trends across high and low responders in terms of patterns of change in cortical activity and type of white matter connectivity. In the long-term, we hope to improve understanding of the process of ADL functional recovery after stroke and optimize robot-training strategies leading to cerebral plasticity. We also hope to determine how lesion characteristics affect changes seen in function, white matter connectivity, and cortical activity. By, accomplishing these aims, we hope to improve upper extremity function after stroke and reduce disability.

ELIGIBILITY:
Inclusion Criteria:

Stroke:

* 30 to 85 years
* Right-handed (evaluated with handedness survey)
* suffered a unilateral ischemic stroke in the motor control area, which resulted in hemiparesis of the arm (confirmed by medical data),
* at least 6-months post-stroke
* residual movement at least (a) 15 degree shoulder flexion or adduction, (b) 15 degree active elbow flexion and extension
* not claustrophobic
* not depressed (as measured depression survey)
* able to use the scanner, i.e., passes the fMRI screening survey
* able to understand the instructions and complete the tracking tasks Control
* older than 20 years
* Right-handed (evaluated with survey)
* not claustrophobic
* able to use the scanner, i.e., passes the fMRI screening survey
* able to understand the instructions and complete the tracking tasks
* no history of neurological disorders --not depressed (as measured depression survey)

Exclusion Criteria:

Stroke:

* brain stem, stroke
* pre-existing neurological or psychiatric disorders
* Spasticity >3 at elbow or fingers on Ashworth
* demonstrated visuospatial, language or attention deficits of a severity that prevents understanding the task
* shoulder pain or joint pain during movements
* synkinetic movements or mirror movements
* decline to participate
* will not comply with full protocol
* pregnant
* allergic to goretex and conductivity gel

Control

* decline to participate
* will not comply with full protocol
* pregnant
* allergic to goretex and conductivity gel

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical Measures: Fugl-Meyer (Motor control), Functional Hand Evaluation (ADL), Jebsen Taylor | Pre (2x) , Post, Follow-Up
Biomechanical:Movement Time, Grasp Aperture, Movement Smoothness | Pre (2x), Post, Follow-up
Imaging Measures: BOLD response (activation), Laterality Index, Fractional Anisotropy, Fiber Density Index | Pre (1x), Post, Follow-up

SECONDARY OUTCOMES:
Clinical Measures: Joint ROM, MMT, Spasticity | Pre(2x), Post, Follow-up
Clinical Measures: Pain, Exertion | During Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michel Torbey, MD, Study Chair — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J Zablocki VA, Milwaukee, Wisconsin